CLINICAL TRIAL: NCT05624697
Title: Assessment of Digital and Clinical Workflow Using Patient Specific Sticky Bone /Implant Housing PEEK Shell in Anterior Atrophic Maxilla: A Case Series
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Samy Bahgat, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16722
Record Dates: First submitted 2022-11-13; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Ridge Augmentation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmented group (Other): Patient Specific Sticky Bone /Implant Housing PEEK Shell in Anterior Atrophic Maxilla with simultaneous implant placement
  Interventions: Procedure: sticky bone housed in PEEK Shell

INTERVENTIONS:
Procedure: sticky bone housed in PEEK Shell — Patient specific Sticky Bone/Implant housing PEEK shell in Anterior Atrophic Maxilla

SUMMARY:
10 Patients having horizontally deficient anterior maxillary areas will be recruited and a preoperative CBCT will be done. The plan is to graft the defective ridges with simultaneously placing dental implants using a PEEK shell that will be specifically designed, constructed and 3D printed to act as a surgical guide for osteotomy drilling and implant placement as well as housing both the implant and the sticky bone (using a mixture of autogenous bone harvested from the symphysis area and xenograft both mixed with plasmatic matrix); that will be added to augment the defective ridge; the PEEK shell will also act as a barrier membrane for Guided Bone Regeneration and will add more stability to the placed implants that will be fixed to the PEEK shell occlusally with a Ti - based abutment.

Primary stability will be measured using Ostell and an immediate postoperative CBCT will be done and superimposed on the preoperative CBCT and an accuracy of plan transfer will be measured to make sure the planning was followed accurately.

Then 6 months later, another CBCT will be done to check the bone gain and quality and a second surgery will be done to remove the PEEK shell and proceed with the conventional implant prosthetic phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Multiple missing Maxillary Anterior Teeth with horizontally defective ridges having adequate soft tissue ample.
* Patients who already gave their consent for this trial.
* Males and females both will be included.

Exclusion Criteria:

* Patients on bisphosphonates or drugs altering bone metabolism, within 2 months before initiating the study.
* Subjected to irradiation in the head and neck region within the last year
* Patients allergic to drugs used in the study like ( Articaine, Lidocaine,
* Patients having a history of a major medical condition (ASA 3,4)
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Active infection or severe inflammation in the area intended for implant placement.
* Unable to open mouth sufficiently to accommodate the surgical tooling.
* Patients participating in other studies, if the present protocol could not be properly followed.
* Referred only for implant placement or unable to attend a 5-year follow-up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-25 (Estimated); Primary Completion 2023-11-25 (Estimated); Study Completion 2024-05-25 (Estimated)

PRIMARY OUTCOMES:
Bone gain | T0 before surgery, T1 immediately after surgery and T2 after 6 months
  Serial CBCT images (T0 before surgery, T1 immediately after surgery and T2 after 6 months) measuring bone gain in mm

SECONDARY OUTCOMES:
Clinically successful osseointegrated implant | At the day of the surgery and 6 months after first surgery
  measuring primary stability immediately after implant placement and in the second surgery using Ostell device
Accuracy of Plan Transfer | 1-3 days postoperatively
  superimposing the preoperative CBCT and the immediately postoperative CBCT to measure the accuracy of the procedure compared to the plan done
Bone Quality | 0 before surgery, T1 immediately after surgery and T2 after 6 months
  Serial CBCT images (T0 before surgery, T1 immediately after surgery and T2 after 6 months) measuring bone quality in Hounsfield units

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt